CLINICAL TRIAL: NCT02369510
Title: Does the Addition of Epinephrine Increase the Duration of Intrathecal Hyperbaric Bupivacaine for Repeat Cesarean Section?
Brief Title: Does the Addition of Epinephrine Prolong the Duration of Spinal Anesthesia for Repeat Cesarean Section?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Assistant Professor of Anesthesiology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GCO 14-2058
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Spinal Anesthesia; Cesarean Section
Keywords: spinal anesthesia; epinephrine; bupivacaine; repeat cesarean
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-dose epinephrine (Experimental): 100micrograms of epinephrine group
  Interventions: Drug: Low-dose epinephrine
- High-dose epinephrine (Experimental): 200micrograms of epinephrine group
  Interventions: Drug: High-dose epinephrine
- No epinephrine (Placebo Comparator): 0.2ml saline
  Interventions: Drug: No epinephrine

INTERVENTIONS:
Drug: Low-dose epinephrine — 0.1ml of preservative-free saline and 0.1ml of 1:1000 epinephrine will be added to the standard spinal medications
  Arms: Low-dose epinephrine
Drug: High-dose epinephrine — 0.2ml of 1:1000 epinephrine will be added to the standard spinal medications
  Other Names: adrenaline
  Arms: High-dose epinephrine
Drug: No epinephrine — 0.2ml of preservative-free saline will be added to the standard spinal medications
  Other Names: preservative-free saline
  Arms: No epinephrine

SUMMARY:
The purpose of this study is to investigate whether the addition of a medication called epinephrine to spinal medications prolongs the duration of the anesthesia. The medication standardly used in spinal anesthesia is a local anesthetic (bupivacaine) and an opiate pain medication (morphine). These medications typically last about 2 hours. The investigators want to determine if adding epinephrine to the spinal medications prolongs the anesthetic without side effects. A longer duration of anesthesia may be useful in prolonged repeat cesarean section. Epinephrine is known to prolong the action of some local anesthetics, but the investigators want to specifically study combining it with the medications the investigators use regularly for cesarean section.

You may qualify to take part in this research study because you are having a repeat cesarean section. Repeat cesarean sections sometimes last longer than 2 hours. The investigators want to determine if epinephrine will prolong the anesthetic.

DETAILED DESCRIPTION:
Spinal anesthesia with bupivacaine is a commonly used anesthetic in the obstetric population. It is most frequently carried out as a single shot intrathecal injection. This method can be utilized for both labor analgesia and surgical anesthesia for cesarean section. One of the concerns in using a single shot spinal injection for surgical anesthesia is the duration of adequate surgical conditions. This concern is especially relevant to repeat cesarean sections, as each subsequent procedure has the potential to be more complex than the prior and, therefore, prolonged. A reliable way to prolong surgical anesthesia provided by single shot spinal injection of bupivacaine could prove invaluable in the setting of repeat cesarean section. It has been well documented that adding epinephrine to intrathecal lidocaine will increase its duration1, but the evidence for augmenting the duration of anesthesia provided by adding epinephrine to bupivacaine is much more equivocal and less robust. This is a randomized control trial investigating whether or not adding epinephrine to a standard single intrathecal injection of hyperbaric bupivacaine for repeat cesarean will prolong its duration. It will be investigated using women who are undergoing scheduled repeat cesarean section in whom neuraxial anesthesia is the appropriate primary anesthetic. The investigators will compare the onset, quality and duration of both sensory and motor components of the spinal block as well as the incidence of known side effects.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent repeat cesarean section
* Neuraxial anesthesia as the planned primary anesthetic
* Informed consent obtained
* Females age 18-50

Exclusion Criteria:

* Emergency cesarean section
* Anesthetic other than neuraxial
* Allergy to local anesthetics, morphine, or epinephrine
* Pre-existing sensory/motor deficit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Yaakov Beilin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Katz D, Hamburger J, Gutman D, Wang R, Lin HM, Marotta M, Zahn J, Beilin Y. The Effect of Adding Subarachnoid Epinephrine to Hyperbaric Bupivacaine and Morphine for Repeat Cesarean Delivery: A Double-Blind Prospective Randomized Control Trial. Anesth Analg. 2018 Jul;127(1):171-178. doi: 10.1213/ANE.0000000000002542. PMID 29077615

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Started | 23 | 22 | 23
Completed | 21 | 19 | 17
Not Completed | 2 | 3 | 6
Not completed — Spilled Medication | 1 | 2 | 1
Not completed — Epidural Activation | 1 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine | Total
Number analyzed (Participants) | 23 | 22 | 23 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (3.86) | 34 (5.19) | 34 (5.12) | 34 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 23 | 68
  Male | 0 | 0 | 0 | 0
Pre-op Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 116 (12) | 119 (10) | 115 (11) | 117 (11)
Pre-op Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 70 (11) | 70 (9) | 66 (8) | 70 (10)
Pre-op Heart Rate (HR) [Mean (Standard Deviation); unit: beats per minute] | 82 (10) | 85 (9) | 78 (10) | 82 (10)

OUTCOME MEASURES:

1. Primary Outcome: Sensory Recovery
Description: Time to T10 sensory recovery as measured by pinprick sensation
Time Frame: up to 3 hours
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 21 | 19 | 17
minutes | 135 [120 to 150] | 165 [150 to 180] | 120 [45 to 150]

2. Secondary Outcome: Motor Recovery
Description: Time to Bromage 3 motor recovery
Time Frame: up to 4 hours
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 21 | 19 | 17
minutes | 150 [135 to 150] | 172 [150 to 210] | 120 [105 to 120]

3. Secondary Outcome: Block Onset
Description: Time to a onset of T4 level of anesthesia or the highest level achieved in 15min
Time Frame: up to 15 min
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 21 | 19 | 17
minutes | 6 [6 to 8] | 8 [6 to 8] | 8 [6 to 10]

4. Secondary Outcome: Number of Participants With Hypotension
Description: Incidence of hypotension as measured by participants needing vasopressor agents
Time Frame: at 2 minutes and at 25 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 21 | 19 | 17
Participants
  2 minutes | 5 | 2 | 8
  25 minutes | 3 | 9 | 3

5. Secondary Outcome: Adequacy of Anesthesia
Description: As measured by pinprick sensation and/or patient discomfort as measured by verbal pain score on a scale of 0=no pain to 10=worst imaginable pain, obtained within 3 hours of receiving anesthesia.
Time Frame: up to 3 hrs
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 21 | 19 | 17
units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 3]

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction score was elicited upon arrival to the recovery room on a 1-5 Likert scale. Number of participants selecting the highest score of 5 or "completely satisfied".
Time Frame: up to 3 hours
Measure: Number; unit: percentage of participants
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 21 | 19 | 17
percentage of participants | 90 | 85 | 87

7. Secondary Outcome: Incidence of Nausea and Vomiting
Time Frame: up to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 21 | 19 | 17
Participants
  2 minutes | 2 | 0 | 4
  25 minutes | 3 | 6 | 1

8. Secondary Outcome: Incidence of Pruritus
Description: data not collected
Time Frame: up to 3 hours
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Low-dose Epinephrine | High-dose Epinephrine | No Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes